CLINICAL TRIAL: NCT01105715
Title: cLDL as a Cardiovascular Disease Risk Factor in Rheumatoid Arthritis
Brief Title: Low Density Lipoprotein Cholesterol (CLDL) as a Cardiovascular Disease Risk Factor in Rheumatoid Arthritis
Acronym: cLDL in RA
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: UAMS 112170
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Disease
Keywords: Rheumatoid Arthritis; cLDL; Cardiovascular disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a subject consents, any blood samples remaining after the tests planned for this study will be stored indefinitely for potential future new studies. Any future new studies using these blood samples will require prior approval by the UAMS Institutional Review Board (IRB). A subject may request destruction of the stored samples at any time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis (RA) Case Subjects: * Fulfill the American College of Rheumatology (ACR) 1987 Classification Criteria for RA
  * Have currently active disease as assessed by Clinical Disease Activity Index (CDAI) score of >10
  * Have > or = 3 swollen joints
- Control Subjects: * Age, sex, and 5-year age categories matched to cases
  * No historical diagnosis of RA and other primary autoimmune or inflammatory disorders

SUMMARY:
The investigators hypothesize that cLDL levels are elevated in RA patients and represents an important mechanism for accelerated atherosclerosis leading to excess cardiovascular disease (CVD) in rheumatoid arthritis (RA) patients. The purpose of this study is to improve understanding of the reasons for increased cardiovascular diseases (such as heart attack and stroke) seen in patients with rheumatoid arthritis (RA, an arthritis that causes inflammation and destruction of joints). Specifically, the study plans to determine whether a particular type of change in proteins in LDL cholesterol ("bad cholesterol") known as carbamylation is an important risk factor for cardiovascular diseases in RA patients. The study will utilize a case-control study design. A total of 120 subjects (males and females between the ages of 18 and 80) may be enrolled in order to ensure that 100 subjects (50 RA case subjects and 50 age and sex matched controls) complete the study. Procedures will consist of a single visit for each subject during which a screening evaluation, an enrollment evaluation, and a single blood draw will be performed.

ELIGIBILITY:
Inclusion Criteria:

For Cases:

* Fulfill the American College of Rheumatology (ACR) 1987 Classification Criteria for RA
* Have currently active disease as assessed by Clinical Disease Activity Index (CDAI)score (a validated composite RA activity index) of > 10
* Have ≥ 3 swollen joints

For Controls:

* Control subjects will be age, sex, and 5-year age categories matched to cases
* No historical diagnosis of RA and other primary autoimmune or inflammatory disorders

Exclusion Criteria:

For both cases and controls:

Renal failure (estimated GFR < 60 ml/min) documented within 3 months of study enrollment (from either subject's self-report or review of available medical records)

* Known clinical history of CVD
* Current cancer (other than skin)
* Current or recent (within past 2 weeks) infection
* Individuals taking lipid-lowering medications
* Any other condition the PI staff feels will jeopardize the health and welfare of the participants
* Rheumatoid vasculitis (for cases only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the UAMS Rheumatology Clinic at the UAMS Outpatient Center, Little Rock, other UAMS outpatient clinics, or through advertisement at the UAMS campus and/or the community.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States